CLINICAL TRIAL: NCT00772031
Title: NINDS Clinical Research Collaboration Chronic Migraine Treatment Trial
Brief Title: NINDS CRC Chronic Migraine Treatment Trial
Acronym: CMTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anne Lindblad (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Anne Lindblad, Executive Vice President, The EMMES Corporation, The Emmes Company, LLC
Organization: The Emmes Company, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-CRC-01; HHSN265200523641C (Other: NINDS Contract)
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Migraine
Keywords: chronic migraine, migraine prevention, chronic headache
MeSH Terms: conditions — Headache Disorders | interventions — Propranolol; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive propranolol and topiramate.
  Interventions: Drug: propranolol LA; Drug: topiramate
- 2 (Placebo Comparator): Participants will receive a placebo and topiramate.
  Interventions: Drug: topiramate; Drug: placebo

INTERVENTIONS:
Drug: propranolol LA — Propranolol LA up to 240 mg/day
  Other Names: Inderal LA
  Arms: 1
Drug: topiramate — Topiramate is an effective, safe and generally well-tolerated drug used for treating chronic migraine. It is becoming the standard treatment among headache specialists.
Drug: placebo — an inactive substance
  Arms: 2

SUMMARY:
The purpose of this study is to compare the reduction in the number of severe headache days at six months in people with chronic migraine treated with topiramate and propranolol versus those treated with topiramate and a placebo.

DETAILED DESCRIPTION:
Chronic migraine affects about 2 percent of all adults. Currently there are no effective preventative treatments to deal with this disabling condition. Three randomized, placebo-controlled trials found that topiramate was an effective, safe and generally well-tolerated drug for treating chronic migraine. As a result of these trials, topiramate is becoming the standard treatment among headache specialists. Experts agree that treatment with combinations of preventive agents is required in the majority of individuals with chronic migraine for maximal headache relief. No randomized trials have assessed the value of frequently used combinations of preventive agents for chronic migraine.

The goal of this trial is to determine if adding a second drug to topiramate treatment will further reduce the headache burden for people with this condition. In the study, 250 participants with chronic migraine will be randomized to two groups - treatment with topiramate and propranolol or topiramate and placebo. Participants will be followed for six months.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic migraine for at least 6 months
* Age ≥ 18 years and age of migraine onset 60 or younger
* EKG performed in the last 12 months

Exclusion Criteria:

* Prior neuro-imaging suggesting secondary structural causes of headache
* Beck Depression Inventory FastScreen score of 13 or greater or other severe psychiatric disorder
* Contraindication to or prior intolerance of topiramate or propranolol (no history of sinus bradycardia, heart block, heart failure, diabetes prone to hypoglycemia, asthma, kidney stones)
* History of kidney failure or nephrolithiasis
* A female who is currently pregnant or lactating or planning to become pregnant in the next year, or is of child-bearing potential and not practicing an acceptable form of birth control
* Currently requires butalbital or opioid drugs for acute headache treatment 10 or more days a month
* Failure of prior trials with at least 50 mg of topiramate combined with at least 80 mg of propranolol
* Use of other migraine preventive drugs (Medications graded as groups 1, 2, 3, and 4 in the AAN Evidence-based Guideline: valproate, divalproex sodium, gabapentin, amitriptyline, nortriptyline, protriptyline, beta-blocker, calcium channel blocker, cyproheptadine; and tizanidine) within the last two months or has received botulinum toxin injection in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Dodick, MD, Principal Investigator — Professor of Neurology, Mayo Clinic; Stephen D. Silberstein, MD, Principal Investigator — Professor of Neurology, Thomas Jefferson University; Deborah Hirtz, MD, Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (39):
- United States (39):
  - Mayo Clinic 5777 E Mayo Blvd, Phoenix, Arizona
  - Paradigm Clinical, Inc. 1324 W. Prince Rd, Tuscon, Arizona
  - Dr. Stephen David Forner - 1405 Magnolia Avenue, Suite B, Chico, California
  - Shanti Clinical Trials, 1880 West Washington Street, Colton, California
  - NervPro Research, 15825 Laguna Canyon Road, Suite 202, Irvine, California
  - Mercy Medical Group- CHWMF 3000 Q Street, Neurology, Sacramento, California
  - Health Sciences America, LLC, 1515 N Federal Hwy, Suite 105, Boca Raton, Florida
  - Southeast Clinical Research, LLC, 304 NE 1st Street, Chiefland, Florida
  - Scientific Clinical Research, Inc 1065 NE 125th Street , Ste 417, Miami, Florida
  - Neurology Associates of Ormond Beach 8 Mirror Lake Drive Suite A&B, Ormond Beach, Florida
  - Neurologique Foundation, Inc. 6 Fairfield Blvd. Suite 11, Ponte Vedra, Florida
  - Neurology Clinical Research, Inc, 3540 North Pine Island Rd, Sunrise, Florida
  - Dr. B. Abraham, P.C. 3020 Highway 124, Snellville, Georgia
  - Ft. Wayne Neurological Center 7956 W. Jefferson Blvd., Fort Wayne, Indiana
  - MidAmerica Neuroscience Research Foundation, 8550 Marshall Dr, Suite 100, Lenexa, Kansas
  - Trover Health System Center for Clinical Studies, 200 Clinic Drive, Madisonville, Kentucky
  - New England Center for Clinical Research (NECCR), 52 Brigham St #7, New Bedford, Massachusetts
  - New England Regional Headache Center, Inc 85 Prescott St, Ste 101, Worcester, Massachusetts
  - ClinSite, LLC 24 Frank Lloyd Wright Drive, Lobby M, Ann Arbor, Michigan
  - Anderson & Collins Clinical Research 1 Ethel Road, Suite 106B, Edison, New Jersey
  - Dent Neurologic Institute, 3980 Sheridan Drive, Amherst, New York
  - Island Neurological Associates, PC, 824 Old Country Road, Plainview, New York
  - Schenectady Neurological Consultants 1401 Union Street, Schenectady, New York
  - Montefiore Headache Center 1575 Blondell Avenue Ste 225, The Bronx, New York
  - Mission Neurology, Research Institute Mission Hospital, 509 Biltmore, Asheville, North Carolina
  - Guilford Neurologic Associates, 1126 North Church Street, Suite 200, Greensboro, North Carolina
  - ClinExcel Research 7908 Cincinnati-Dayton Rd, Ste J, West Chester, Ohio
  - Abington Neurological Associates, Ltd., 1245 Highland Avenue, Ste 301, Abington, Pennsylvania
  - Neurology and Sleep Medicine PC, 701 Ostrum Street, Suite 302, Bethlehem, Pennsylvania
  - Jefferson Headache Center/Thomas Jefferson Univ. 111 South 11th Street, Suite 8130, Philadelphia, Pennsylvania
  - Progress Clinical Trials, 707 Kings Lane, Tullahoma, Tennessee
  - Texas Neurology, PA, 6301 Gaston Avenue, Suite 400 West Tower, Dallas, Texas
  - Houston Headache Clinic, 1213 Hermann Drive, Suite 820, Houston, Texas
  - Houston Sleep Center, Todd J. Swick, MD, PA, 7500 San Felipe, Suite 525, Houston, Texas
  - Protenium Clinical Research, LLC 1725 Chadwick Court Suite 200, Hurst, Texas
  - Starlight Clinical Research, 1325 W. South Jordan Pkwy, Ste 101, South Jordan, Utah
  - Swedish Pain & Headache Center 101 Madison St, Suite 200, Seattle, Washington
  - West Virginia University 1 Medical Center Dr, Box 9180, Morgantown, West Virginia
  - Gundersen Clinic, Ltd, 1836 South Avenue, MS: EB3-002, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate Plus Propranolol: Participants will receive propranolol and topiramate.
- Topiramate Plus Placebo: Participants will receive a placebo and topiramate.
Period: Overall Study
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Started | 96 | 95
Completed | 64 | 52
Not Completed | 32 | 43
Not completed — Early termination of trial | 12 | 10
Not completed — Lost to Follow-up | 20 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo | Total
Number analyzed (Participants) | 96 | 95 | 191
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 94 | 92 | 186
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 39.8 (1.09) | 41.2 (1.15) | 40.5 (0.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 88 | 172
  Male | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 96 | 95 | 191

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Moderate to Severe Headache Days Within a 28 Day Average Period in Six Months Compared to Baseline
Description: (Number of moderate to severe headache days (as defined by the International Headache Society Guidelines (2006)) counted over a 28 day diary period at baseline (before treatment with propranolol or placebo)) minus (the number of moderate to severe headache days counted over a 56 day diary period (weeks 16-24 post treatment) divided by 2).
Time Frame: Baseline (pre-randomization), months 5 and 6 post randomization
Population: ITT to the extent diary information was available. Available defined as all subjects with 12 or more diary entries between 16 and 24 weeks. Multiple imputation used on all randomized subjects as a sensitivity analysis on the primary outcome.
Measure: Mean (Standard Deviation); unit: Moderate to severe headache days
Groups:
- Topiramate Plus Placebo: Participants will receive placebo and topiramate.
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Number analyzed (Participants) | 63 | 48
Moderate to severe headache days | 4.4 (5.98) | 4.7 (5.66)
Statistical Analysis 1: Comparison: Topiramate Plus Propranolol vs Topiramate Plus Placebo; The study was designed to enroll 250 subjects to provide at least 90% power to detect a 3-day difference and 87% power to detect a 2.5-day difference in 28-day moderate-to-severe headache rate reductions at six months, assuming a type I error rate of 0.05, a two-sided test, a 10% loss to follow-up and a standard deviation of within-person change in days with headache of six; Test type: Superiority or Other; p = 0.77, ANCOVA; covariate adjustments: study site, baseline mod-to-sev 28-day headache-rate, topiramate use, medication overuse, and anti-depressive medications use; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.8 to 2.4], Standard Error of Mean 0.97 — Topiramate plus placebo mean reduction minus topiramate plus propranolol reduction

2. Secondary Outcome: Number of Subjects Experiencing at Least a 30% Reduction in 28-day Moderate to Severe Headache Days
Time Frame: 6 months post randomization
Population: All subjects randomized with opportunity for 6 month followup. Due to early study termination those who did not have opportunity for 6 month followup at time of study closure were excluded. All lost to followups were counted as failure
Measure: Number; unit: participants
Groups:
- Topiramate Plus Proporanolol: Participants will receive propranolol and topiramate.
Arm/Group | Topiramate Plus Proporanolol | Topiramate Plus Placebo
Number analyzed (Participants) | 84 | 82
participants | 37 | 28
Statistical Analysis 1: Comparison: Topiramate Plus Proporanolol vs Topiramate Plus Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.75 to 2.78]

3. Secondary Outcome: Number of Subjects Experiencing at Least a 50% Reduction in 28-day Moderate to Severe Headache Days
Time Frame: 6 months
Population: All participants with the opportunity for 6-month follow-up. Due to early study termination some participants were randomized and did not have the opportunity to be followed for six months
Measure: Number; unit: participants
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Number analyzed (Participants) | 84 | 82
participants | 26 | 23
Statistical Analysis 1: Comparison: Topiramate Plus Propranolol vs Topiramate Plus Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 1.00, 95% CI [0.50 to 2.02]

4. Secondary Outcome: Change From Baseline in Beck's Depression Inventory FastScreen Score at 6 Months
Description: Total score from Beck's Depression Inventory FastScreen at 6 months minus total score from Beck's Depression Inventory FastScreen at baseline. Scale scores range from 0 to 21 with higher values indicating worsening depression. the following categories separate participants into groups of depression levels: Minimal (Score 0-3), Mild (Score 4-8),Moderate (Score 9-12),Severe (Score 13-21).
Time Frame: Baseline and 6 months
Population: The number who completed the Beck's Depression Inventory at baseline and three months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Number analyzed (Participants) | 53 | 44
units on a scale | 0.3 (0.25) | 0.6 (0.30)

5. Secondary Outcome: Change From Baseline in Migraine Disability Assessment (MIDAS) Score at 6 Months
Description: MIDAS scoring ranges from 0 to 270. The scores are divided into ranges of disability with higher scores indicating increased disability as follows: 0-5 (Grade I - Minimal or infrequent disability); 6-10 (Grade II - Mild or infrequent disability); 11-20 (Grade III - Moderate disability); and 21+ (Grade IV - Severe disability).
Time Frame: Baseline and 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Number analyzed (Participants) | 53 | 44
units on a scale | -3.18 (3.70) | -3.46 (3.82)
Statistical Analysis 1: Comparison: Topiramate Plus Propranolol vs Topiramate Plus Placebo; Test type: Superiority or Other; p = 0.91, ANCOVA; Mean Difference (Net) = -0.28, Standard Deviation 3.75

6. Secondary Outcome: Change From Baseline in Migraine Specific Quality of Life (MSQ)-Role Restrictive Score at 6 Months
Description: The MSQ (version 2.1 copyrighted 1992, 1996, 1998 by Glaxo Wellcome Inc., Research Triangle Park, North Carolina) is a 14 item questionnaire. Item responses are summed and scored as a total score and three domains: Role Preventive, Role Restrictive, Emotional Function. Scores within each domain are rescaled to range from 0 to 100. A lower score indicates a poorer quality of life associated with that domain or in total. Because of the observed interaction within a domain, only domain scores were used as outcome measures for this study.
Time Frame: baseline and 6 months post randomization
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Number analyzed (Participants) | 53 | 62
units on a scale | -0.7 (5.5) | -2.2 (5.71)

7. Secondary Outcome: Change From Baseline in Migraine-Specific Quality of Life (MSQ)-Role Preventive at 6 Months
Description: as for outcome 6
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Topiramate Plus Propranolol, no Prior, Stable Topiramate: Participants without prior stable topiramate use received propranolol and topiramate.
- Topiramate Plus Placebo, no Prior, Stable Topiramate: Participants without prior stable topiramate use received a placebo and topiramate.
- Topiramate Plus Propranolol, Prior, Stable Topiramate: Participants with prior stable topiramate use received propranolol and topiramate.
- Topiramate Plus Placebo, Prior, Stable Topiramate: Participants with prior stable topiramate use received a placebo and topiramate.
Arm/Group | Topiramate Plus Propranolol, no Prior, Stable Topiramate | Topiramate Plus Placebo, no Prior, Stable Topiramate | Topiramate Plus Propranolol, Prior, Stable Topiramate | Topiramate Plus Placebo, Prior, Stable Topiramate
Number analyzed (Participants) | 40 | 31 | 13 | 13
units on a scale | 12.9 (2.88) | 5.9 (3.10) | -11.5 (5.00) | 11.0 (5.06)

8. Secondary Outcome: Change From Baseline in Migraine-Specific Quality of Life (MSQ) - Emotional Function at 6 Months
Description: as for outcome 6
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Number analyzed (Participants) | 53 | 62
units on a scale | 8.9 (3.43) | 9.8 (3.80)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Self report and systematic questions at scheduled visits(Tingling or prickling;Nausea/Vomiting;Weight loss;Weight gain;More than usual fatigue;Depression;Trouble thinking;New or unusual problems with memory;Racing, pounding or skipping of heart(more than 1 time);Dizziness(more than 1 time);Impotence).
Arm/Group | Topiramate Plus Propranolol | Topiramate Plus Placebo
Serious Adverse Events (participants affected / at risk) | 7/96 | 5/95
Other Adverse Events (participants affected / at risk) | 59/96 | 50/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate Plus Propranolol (N=96) | Topiramate Plus Placebo (N=95)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Upper Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Colporrhaphy (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate Plus Propranolol (N=96) | Topiramate Plus Placebo (N=95)
Dizziness (Nervous system disorders) | 13 | 3
Memory Impairment (Nervous system disorders) | 6 | 8
Mental Impairment (Nervous system disorders) | 12 | 7
Paraesthesia (Nervous system disorders) | 12 | 10
Depression (Psychiatric disorders) | 8 | 3
Insomnia (Psychiatric disorders) | 2 | 7
Fatigue (General disorders) | 22 | 11
Any Vascular Disorder (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less